CLINICAL TRIAL: NCT03448393
Title: Phase 1 Dose Escalation Study of CD19/CD22 Chimeric Antigen Receptor (CAR) T Cells in Children and Young Adults With Recurrent or Refractory CD19/CD22-expressing B Cell Malignancies
Brief Title: CD19/CD22 Chimeric Antigen Receptor (CAR) T Cells in Children and Young Adults With Recurrent or Refractory CD19/CD22-expressing B Cell Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Nirali N. Shah, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 180059; 18-C-0059
Record Dates: First submitted 2018-02-27; First posted 2018-02-28 (Actual); Results first posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, B Cell; B-Cell Lymphoma; B-Cell Leukemia; Acute Lymphoid Leukemia; B-Non Hodgkin Lymphoma; B-NHL; B-All; Acute Lymphoblastic Leukemia; Acute Lymphocytic Leukemia
Keywords: B-Non Hodgkin Lymphoma; Acute Lymphocytic Leukemia; Acute Lymphoblastic Leukemia; B-precursor ALL; B-All; Philadelphia chromosome + ALL; Lymphoma; CD-22 Expressing Tumor; CD-19 expressing tumor; Adoptive Immunotherapy
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, B-Cell; Lymphoma, B-Cell; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Philadelphia Chromosome; Lymphoma | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; Blood Component Removal; Antiemetics; Diphenhydramine; Acetaminophen; Electrocardiography; Echocardiography; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): Cluster of differentiation 19 (CD19)/cluster of differentiation 22 (CD22)-chimeric antigen receptor (CAR)-transduced T cells at escalating doses.
  Interventions: Biological: CD19/CD22 CAR T-Cells; Drug: Fludarabine; Drug: Cyclophosphamide; Procedure: Apheresis; Other: Anti-emetic; Drug: Diphenhydramine; Drug: Acetaminophen; Diagnostic Test: ECG; Diagnostic Test: ECHO; Diagnostic Test: MRI Brain; Procedure: Bone marrow biopsy; Diagnostic Test: Cardiac MRI
- Dose Expansion (Experimental): Cluster of differentiation 19 (CD19)/cluster of differentiation 22 (CD22)-chimeric antigen receptor (CAR)-transduced T cells at maximum tolerated dose (MTD) or highest dose administered.
  Interventions: Biological: CD19/CD22 CAR T-Cells; Drug: Fludarabine; Drug: Cyclophosphamide; Procedure: Apheresis; Other: Anti-emetic; Drug: Diphenhydramine; Drug: Acetaminophen; Diagnostic Test: ECG; Diagnostic Test: ECHO; Diagnostic Test: MRI Brain; Procedure: Bone marrow biopsy; Diagnostic Test: Cardiac MRI

INTERVENTIONS:
Biological: CD19/CD22 CAR T-Cells — Cluster of differentiation 19 (CD19)/cluster of differentiation 22 (CD22) chimeric antigen receptor (CAR) T-cells will be infused on Day 0 after lymphodepleting chemotherapy regimen.
  Other Names: cluster of differentiation 19 chimeric antigen receptor T-cells; cluster of differentiation 22 chimeric antigen receptor T-cells
Drug: Fludarabine — Fludarabine is administered as an intravenous (IV) infusion in an appropriate solution over 30 minutes. To prevent undue toxicity the dose will be based on body surface area (BSA) (25-30 mg/m^2/dose) on Days -4, -3, -2 or Days -5, -4, -3, -2.
  Other Names: Fludara
Drug: Cyclophosphamide — Cyclophosphamide will be diluted in an appropriate solution and infused over one hour. The dose will be based on the body surface area (BSA), at 900 mg/m^2/dose after fludarabine infusion on Day -2 or 600 mg/m^2/dose on Days -3 & -2.
  Other Names: Cytoxan
Procedure: Apheresis — According to institutional standards.
Other: Anti-emetic — Prophylaxis and treatment.
Drug: Diphenhydramine — Pre-medication: 0.5-1 mg/kg/dose (maximum 50 mg/dose) by mouth or intravenous over 10-15 minutes.
  Other Names: Benadryl; Banophen; Nytol
Drug: Acetaminophen — Pre-medication: 15 mg/kg/dose (maximum 650 mg/dose by mouth).
  Other Names: Tylenol; ofirmev; FeverAll
Diagnostic Test: ECG — Pre-cell infusion.
  Other Names: Electrocardiogram
Diagnostic Test: ECHO — Pre-cell infusion.
  Other Names: Echocardiogram
Diagnostic Test: MRI Brain — Pre-cell infusion.
  Other Names: Magnetic resonance imaging
Procedure: Bone marrow biopsy — Pre-cell infusion.
  Other Names: BM biopsy
Diagnostic Test: Cardiac MRI — Screening
  Other Names: Cardiac magnetic resonance imaging

SUMMARY:
Background:

B-cell leukemias and lymphomas are cancers that are often difficult to treat. The primary objective of this study is to determine the ability to take a patient's own cells (T lymphocytes) and grow them in the laboratory with the cluster of differentiation 19 (CD19/cluster of differentiation 22-chimeric antigen receptor (CD22-CAR) gene through a process called 'lentiviral transduction (also considered gene therapy) and growing them to large numbers to use as a treatment for hematologic cancers in children and young adults.. Researchers want to see if giving modified CD19/CD22-CAR T cells to people with these cancers can attack cancer cells. In addition, the safety of giving these gene modified cells to humans will be tested at different cell doses. Additional objectives are to determine if this therapy can cause regression of B cell cancers and to measure if the gene modified cells survive in patients' blood.

Objective:

To study the safety and effects of giving CD19/CD22-CAR T cells to children and young adults with B-cell cancer.

Eligibility:

People ages 3-39 with certain cancers that have not been cured by standard therapy. Their cancer tissue must express the CD19 protein.

Design:

A sample of participants blood or bone marrow will be sent to National Institutes of Health (NIH) and tested for leukemia.

Participants will be screened with:

Medical history

Physical exam

Urine and blood tests (including for human immunodeficiency virus (HIV)

Heart and eye tests

Neurologic assessment and symptom checklist.

Scans, bone marrow biopsy, and/or spinal tap

Some participants will have lung tests.

Participants will repeat these tests throughout the study and follow-up.

Participants will have leukapheresis. Blood will be drawn from a plastic tube (intravenous (IV) or needle in one arm then go through a machine that removes lymphocytes. The remaining blood will be returned to the participant's other arm.

Participants will stay in the hospital about 2 weeks. There they will get:

Two chemotherapy drugs by IV

Their changed cells by IV

Standard drugs for side effects

Participants will have frequent follow-up visits for 1 year, then 5 visits for the next 4 years. Then they will answer questions and have blood tests every year for 15 years.

...

DETAILED DESCRIPTION:
Background:

* Acute lymphoblastic leukemia (ALL) accounts for approximately 25% of childhood cancer. Survival rates have improved, but outcomes for some subgroups, including infants and young adults remain poor, and survival for patients who relapse is < 50%, despite allogeneic stem cell transplant following second remission.
* Cluster of differentiation 19 (CD19 immune escape has been observed by several groups following CD19-chimeric antigen receptor (CAR) therapy for B-ALL. Investigation of this phenomenon reveals a complex biology responsible for loss or downregulation of CD19 expression observed in these cases.
* Sequential therapy using cluster of differentiation 22 (CD22)-CARs to treat CD19 dim/lo escape is associated with rapid development of resistance due to CD22 downregulation. This trial will test whether simultaneous targeting of CD19 and CD22 using a novel bivalent CD19/22-CAR is safe and feasible.

Objectives:

-Assess the safety of administering escalating doses of autologous CD19/CD22-CAR engineered T cells that meet established release specifications in children and young adults with CD19+CD22+ B cell ALL, isolated central nervous system (CNS) ALL, or lymphoma following a cyclophosphamide/fludarabine conditioning regimen.

Eligibility:

-Participants between >= 3 years and <= 39 years of age, with CD19+/CD22+ B cell ALL, isolated CNS ALL, or lymphoma who have relapsed or have refractory disease after at least one standard chemotherapy regimen and one salvage regimen, with no alternative curative options who meet standard Phase I eligibility criteria.

Design:

* Phase I, 3 + 3 dose escalation design using the following dose levels: -1: 1 x 10^5 transduced T cells/kg (+/- 20%); 1: 3 x 10^5 transduced T cells/kg (+/- 20%); 2: 1 x 10^6 transduced T cells/kg; and 3: 3 x 10^6 transduced T cells/kg (+/- 20%); 4: 1 x 10^7 transduced T cells/kg (+/- 20%).
* Participants will receive a lymphodepleting preparative regimen of fludarabine (25 mg/m^2/day (d) x 3 on Days -4, -3, -2) and cyclophosphamide (900 mg/m^2/d x 1 on Day -2) followed by infusion of CD19/CD22-CAR T-cells on D0. Participants who are CAR pretreated (with exception for those with an interval hematopoietic stem cell transplantation (HSCT) will receive increased lymphodepleting preparative regimen of fludarabine (30^mg/m^2/d x 4 on Days -5, -4, -3, -2) and cyclophosphamide (600 mg/m^2/d x 2 on Days -3, -2) followed by infusion of CD19/CD22-CAR T-cells on D0. If fludarabine is unavailable, pentostatin may be given as an alternative.
* Patients will be evaluated sequentially for toxicity, antitumor effects, CAR expansion and persistence, as well as research correlatives.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

Study subjects with cluster of differentiation 19 (CD19) + cluster of differentiation 22 (CD22+) expressing B cell malignancies who have relapsed or are treatment refractory may enroll as defined by the following inclusion and exclusion criteria.

INCLUSION CRITERIA:

* Diagnosis

  * Participant must have a B cell acute lymphoblastic leukemia (ALL) (inclusive of chronic myeloid leukemia (CML) with ALL transformation) or lymphoma and must have relapsed or refractory disease after at least one standard chemotherapy regimen and one salvage regimen. In view of the principal investigator (PI) and the primary oncologist, there must be no available alternative curative therapies and subjects must be either ineligible for allogeneic stem cell transplant (SCT), have refused SCT, recurred after SCT, or have disease activity that prohibits SCT at the time of enrollment. Participants who have undergone autologous SCT will be eligible, and participants that have undergone allogeneic SCT will be eligible if, in addition to meeting other eligibility criteria, they have no evidence of graft versus host disease (GVHD) and have been without immunosuppressive agents for at least 30 days. Participants with Philadelphia chromosome + ALL must have failed prior tyrosine kinase inhibitor.
  * Participants must have measurable or evaluable disease at the time of enrollment, which may include any evidence of disease including minimal residual disease detected by flow cytometry, cytogenetics, or polymerase chain reaction (PCR) analysis. For those being considered for reinfusions, measurable or evaluable disease is not required at the time of reinfusion.
* CD22/CD19 expression

  --CD19 expression must be detected on greater than 15% of the malignant cells by immunohistochemistry or greater than 90% by flow cytometry. The choice of whether to use flow cytometry or immunohistochemistry will be determined by what is the most easily available tissue sample in each participant. In general, immunohistochemistry will be used for lymph node biopsies, flow cytometry will be used for peripheral blood and bone marrow samples. CD22+ B cell malignancy is required and CD22 expression levels will be documented when available, but a specific level of expression is not an eligibility requirement; it may be documented as positive or negative.
* Age:

  --Greater than or equal to 3 years of age (and at least 15 kg) and less than or equal to 39 years of age at time of enrollment (greater than or equal to 3 years to less than or equal to 39 years). NOTE: The first participant in each dose cohort must be greater than or equal to 18 years of age.
* Clinical Performance

  --Clinical performance status: Participants greater than or equal to 16 years of age: Karnofsky greater than or equal to 50%; Participants < 16 years of age: Lansky scale greater than or equal to 50%. Subjects who are unable to walk because of paralysis, but who are upright in a wheelchair will be considered ambulatory for the purpose of calculating the performance score.
* Participants must have adequate organ and marrow function as defined below:

  * leukocytes greater than or equal to 750/mcL*
  * platelets greater than or equal to 50,000/mcL*
  * total bilirubin less than or equal to 2 X upper limit of normal (ULN) (except in the case of subjects with documented Gilbert's disease > 3x ULN)
  * Aspartate aminotransferase (AST)serum glutamic-oxaloacetic transaminase (SGOT)/alanine aminotransferase (ALT)serum glutamate pyruvate transaminase (SGPT) less than or equal to 10 X institutional upper limit of normal
  * creatinine less than or equal to the maximum for age listed in the table below
  * Age (Years): less than or equal to 5. Maximum Serum Creatinine (mg/dL): less than or equal to 0.8
  * Age (Years): 6 to less than or equal to 10. Maximum Serum Creatinine (mg/dL): less than or equal to 1.0
  * Age (Years): >10. Maximum Serum Creatinine (mg/dL): less than or equal to 1.2
  * OR
  * creatinine clearance greater than or equal to 60 mL/min/1.73 m^2 for participants with creatinine levels above institutional normal.

    * if these cytopenias are not judged by the investigator to be due to underlying disease (i.e. potentially reversible with anti-neoplastic therapy); A subject will not be excluded because of pancytopenia greater than or equal to Grade 3 if it is due to disease, based on the results of bone marrow studies.
* Subjects with central nervous system (CNS) disease are eligible, with exceptions as noted in the exclusion criteria
* Contraception:

  --Individuals of child-bearing or child-fathering potential (IOCBP or IOCFP) must be willing to practice birth control from the time of enrollment on this study and for 12 months after receiving the preparative regimen for IOCBP and for 4 months after receiving the preparative regimen for IOCFP
* Cardiac function: Left ventricular ejection fraction greater than or equal to 45% or fractional shortening greater than or equal to 28%, and no clinically significant electrocardiogram (ECG) findings
* Pulmonary Function
* Baseline oxygen saturation >92% on room air at rest
* Participants with respiratory symptoms must have a diffusing capacity for carbon monoxide (DLCO)/adjusted > 45%. For children who are unable to cooperate for pulmonary function tests (PFTs) they must not have dyspnea at rest or known requirement for supplemental oxygen.
* Ability of subject, parent(s)/guardian(s), Legally Authorized Representative (LAR) or Durable Power of Attorney (DPA) to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

Subjects meeting any of the following criteria are not eligible for participation in the study:

* Recurrent or refractory ALL limited to isolated testicular.
* Subjects with radiologically detected active CNS lymphoma or isolated CNS disease which are eligible for definitive CNS directed radiation therapy will be excluded.
* Hyperleukocytosis (greater than or equal to 50,000 blasts/micro L) or rapidly progressive disease that in the estimation of the investigator and sponsor would compromise ability to complete study therapy;
* Pregnant or nursing individuals.
* Subjects will be excluded related to the following prior therapy criteria:

  * Systemic chemotherapy, anti-neoplastic investigational agents, or antibody-based therapies =<2 weeks (6 weeks for clofarabine or nitrosoureas) prior to apheresis with the following exception:

    ---No time restriction with prior intrathecal chemotherapy, steroid therapy, hydroxyurea or ALL maintenance type chemotherapy (vincristine, 6-mercaptopurine, oral methotrexate, or a tyrosine kinase inhibitor for participants with Philadelphia chromosome (Ph)+ ALL) provided there is recovery from any acute toxic effects.
  * Radiation therapy =<3 weeks prior to apheresis with the following exception:

    ---No time restriction with radiation therapy if the volume of bone marrow treated is less than 10% and the subject has measurable/evaluable disease outside the radiation window.
  * History of allogeneic stem cell transplantation prior to apheresis that meet the following criteria:

    * Less than 100 days post-transplant
    * Evidence of active graft-versus-host disease (GVHD)
    * Taking immunosuppressive agents within 30 days prior to apheresis
    * Less than 6 weeks post donor lymphocyte infusion (DLI)
  * History of prior CAR therapy or other adoptive cell therapies prior to apheresis that meet the following criteria:

    * Less than 30 days post-infusion
    * Circulating CAR T cells (or genetically modified cells) >5% by flow cytometry in peripheral blood.
* Human Immunodeficiency Virus (HIV)/hepatitis B virus (HBV)/hepatitis C virus (HCV) Infection:

  * a. Seropositive for HIV antibody. (Participants with HIV are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy in the future should study results indicate effectiveness.)
  * b. Positive for Hepatitis B surface antigen (HbsAG).
  * c. Evidence of active Hepatitis C (evidenced by detectable HCV ribonucleic acid (RNA)
* Uncontrolled, symptomatic, intercurrent illness including but not limited to infection, congestive heart failure, unstable angina pectoris, cardiac arrhythmia, psychiatric illness, or social situations that would limit compliance with study requirements or in the opinion of the PI would pose an unacceptable risk to the subject;
* Second malignancy other than in situ carcinoma of the cervix, unless the tumor was treated with curative intent at least two years previously and subject is in remission;
* History of severe, immediate hypersensitivity reaction attributed to compounds of similar chemical or biologic composition to any agents used in study or in the manufacturing of the cells.

Ages: 3 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2025-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nirali N Shah, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).

REFERENCES:
- [Derived] Silbert SK, Madan S, Holland EM, Steinberg SM, Little L, Foley T, Epstein M, Sarkisian A, Lee DW, Nikitina E, Kakumanu S, Ruppin E, Shalabi H, Yates B, Shah NN. A comprehensive analysis of adverse events in the first 30 days of phase 1 pediatric CAR T-cell trials. Blood Adv. 2023 Sep 26;7(18):5566-5578. doi: 10.1182/bloodadvances.2023009789. PMID 37486616
- [Derived] Shalabi H, Qin H, Su A, Yates B, Wolters PL, Steinberg SM, Ligon JA, Silbert S, DeDe K, Benzaoui M, Goldberg S, Achar S, Schneider D, Shahani SA, Little L, Foley T, Molina JC, Panch S, Mackall CL, Lee DW, Chien CD, Pouzolles M, Ahlman M, Yuan CM, Wang HW, Wang Y, Inglefield J, Toledo-Tamula MA, Martin S, Highfill SL, Altan-Bonnet G, Stroncek D, Fry TJ, Taylor N, Shah NN. CD19/22 CAR T cells in children and young adults with B-ALL: phase 1 results and development of a novel bicistronic CAR. Blood. 2022 Aug 4;140(5):451-463. doi: 10.1182/blood.2022015795. PMID 35605184
- [Derived] Singh N. Modified T cells as therapeutic agents. Hematology Am Soc Hematol Educ Program. 2021 Dec 10;2021(1):296-302. doi: 10.1182/hematology.2021000262. PMID 34889384
- [Derived] Molina JC, Steinberg SM, Yates B, Lee DW, Little L, Mackall CL, Shalabi H, Shah NN. Factors Impacting Overall and Event-Free Survival following Post-Chimeric Antigen Receptor T Cell Consolidative Hematopoietic Stem Cell Transplantation. Transplant Cell Ther. 2022 Jan;28(1):31.e1-31.e9. doi: 10.1016/j.jtct.2021.10.011. Epub 2021 Oct 20. PMID 34687939
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-C-0059.html

RESULTS

PARTICIPANT FLOW:
Groups:
- GROUP 1: Cohort 1, Dose Level 1, 3 x10^5 Transduced T Cells/kg (+Or-20%): Lymphodepleting chemotherapy regimen with Fludarabine and Cyclophosphamide.
  Fludarabine: Fludarabine is administered as an intravenous (IV) infusion in an appropriate solution over 30 minutes. The dose will be based on body surface area (BSA) at 25 mg/m^2/dose on Day -4, -3, -2.
  Cyclophosphamide: Cyclophosphamide will be diluted in an appropriate solution and infused over one hour. The dose will be based on the body surface area (BSA) at 900 mg/m^2/dose after fludarabine infusion on Day -2.
  Cluster of differentiation 19 (CD19)/cluster of differentiation 22 (CD22)-chimeric antigen receptor (CAR)-transduced T cells Dose Level 1, 3 x10^5 transduced T cells/kg (+or-20%) infused on Day 0 after lymphodepleting chemotherapy regimen
- GROUP 2: Cohort 1, Dose Level 2, 1x10^6 Transduced T Cells/kg (+Or-20%): Lymphodepleting chemotherapy regimen with Fludarabine and Cyclophosphamide.
  Fludarabine: Fludarabine is administered as an intravenous (IV) infusion in an appropriate solution over 30 minutes. The dose will be based on body surface area (BSA) at 25 mg/m^2/dose on Day -4, -3, -2.
  Cyclophosphamide: Cyclophosphamide will be diluted in an appropriate solution and infused over one hour. The dose will be based on the body surface area (BSA) at 900 mg/m^2/dose after fludarabine infusion on Day -2.
  Cluster of differentiation 19 (CD19)/cluster of differentiation 22 (CD22)-chimeric antigen receptor (CAR)-transduced T cells at Dose Level 2, 1x10^6 transduced T cells/kg (+or-20%) infused on Day 0 after lymphodepleting chemotherapy regimen.
- GROUP 3: Cohort 1, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%): Lymphodepleting chemotherapy regimen with Fludarabine and Cyclophosphamide.
  Fludarabine: Fludarabine is administered as an intravenous (IV) infusion in an appropriate solution over 30 minutes. The dose will be based on body surface area (BSA) at 25 mg/m^2/dose on Day -4, -3, -2.
  Cyclophosphamide: Cyclophosphamide will be diluted in an appropriate solution and infused over one hour. The dose will be based on the body surface area (BSA) at 900 mg/m^2/dose after fludarabine infusion on Day -2.
  Cluster of differentiation 19 (CD19)/cluster of differentiation 22 (CD22)-chimeric antigen receptor (CAR)-transduced T cells at Dose Level 3, 3 x10^6 transduced T cells/kg (+or-20%) infused on Day 0 after lymphodepleting chemotherapy regimen
- GROUP 4: Cohort 1A, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%); GROUP 6: Cohort 2A, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%): Participants who are chimeric antigen receptor (CAR) naïve or CAR pre-treated and received an interval transplant.
  Lymphodepleting chemotherapy regimen with Fludarabine and Cyclophosphamide.
  Fludarabine: Fludarabine is administered as an intravenous (IV) infusion in an appropriate solution over 30 minutes. The dose will be based on body surface area (BSA) at 25 mg/m^2/dose on Day -4, -3, -2.
  Cyclophosphamide: Cyclophosphamide will be diluted in an appropriate solution and infused over one hour. The dose will be based on the body surface area (BSA) at 900 mg/m^2/dose after fludarabine infusion on Day -2.
  Cluster of differentiation 19 (CD19)/cluster of differentiation 22 (CD22)-chimeric antigen receptor (CAR)-transduced T cells at Dose Level 3, 3 x10^6 transduced T cells/kg (+or-20%) infused on Day 0 after lymphodepleting chemotherapy regimen
- GROUP 5: Cohort 1B, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%); GROUP 7: Cohort 2B, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%: Participants who previously received Chimeric Antigen Receptor (CAR) therapy. Lymphodepleting chemotherapy regimen with Fludarabine and Cyclophosphamide.
  Fludarabine: Fludarabine is administered as an intravenous (IV) infusion in an appropriate solution over 30 minutes. The dose will be based on body surface area (BSA) at 30 mg/m^2/dose on Day -5, -4, -3, -2.
  Cyclophosphamide: Cyclophosphamide will be diluted in an appropriate solution and infused over one hour. The dose will be based on the body surface area (BSA) at 600 mg/m^2/dose after fludarabine infusion on Day -3 & -2.
  Cluster of differentiation 19 (CD19)/cluster of differentiation 22 (CD22)-chimeric antigen receptor (CAR)-transduced T cells at Dose Level 3, 3 x10^6 transduced T cells/kg (+or-20%) infused on Day 0 after lymphodepleting chemotherapy regimen.
- GROUP 8: Cohort 2C, Dose Level 3, 3 x 10^6 Transduced T-cells/kg (+Or- 20%): Participants with isolated central nervous system (CNS) disease.
  Lymphodepleting chemotherapy regimen with Fludarabine and Cyclophosphamide.
  Fludarabine: Fludarabine is administered as an intravenous (IV) infusion in an appropriate solution over 30 minutes. The dose will be based on body surface area (BSA) at 25 mg/m^2/dose on Day -4, -3, -2.
  Cyclophosphamide: Cyclophosphamide will be diluted in an appropriate solution and infused over one hour. The dose will be based on the body surface area (BSA) at 900 mg/m^2/dose after fludarabine infusion on Day -2.
  Cluster of differentiation 19 (CD19)/cluster of differentiation 22 (CD22)-chimeric antigen receptor (CAR)-transduced T cells at Dose Level 3, 3 x10^6 transduced T cells/kg (+or-20%) infused on Day 0 after lymphodepleting chemotherapy regimen.
- Enrolled and Not Assigned to a Treatment Assignment Code; Not Treated: Participants were enrolled for screening but were not enrolled on treatment.
Period: Dose Escalation
Arm/Group | GROUP 1: Cohort 1, Dose Level 1, 3 x10^5 Transduced T Cells/kg (+Or-20%) | GROUP 2: Cohort 1, Dose Level 2, 1x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 3: Cohort 1, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 4: Cohort 1A, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 5: Cohort 1B, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 6: Cohort 2A, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 7: Cohort 2B, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20% | GROUP 8: Cohort 2C, Dose Level 3, 3 x 10^6 Transduced T-cells/kg (+Or- 20%) | Enrolled and Not Assigned to a Treatment Assignment Code; Not Treated
Started | 4 | 4 | 5 | 2 | 1 | 0 | 0 | 0 | 8
Completed | 4 | 4 | 4 | 2 | 1 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 8
Not completed — Not Treated - participant did not receive cell infusion. | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 8
Period: Dose Expansion
Arm/Group | GROUP 1: Cohort 1, Dose Level 1, 3 x10^5 Transduced T Cells/kg (+Or-20%) | GROUP 2: Cohort 1, Dose Level 2, 1x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 3: Cohort 1, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 4: Cohort 1A, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 5: Cohort 1B, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 6: Cohort 2A, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 7: Cohort 2B, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20% | GROUP 8: Cohort 2C, Dose Level 3, 3 x 10^6 Transduced T-cells/kg (+Or- 20%) | Enrolled and Not Assigned to a Treatment Assignment Code; Not Treated
Started | 0 | 0 | 0 | 0 | 0 | 21 | 1 | 1 | 7
Completed | 0 | 0 | 0 | 0 | 0 | 21 | 1 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7
Not completed — Not treated - screen failure | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7

BASELINE CHARACTERISTICS:
Population: Data collected for participants enrolled and not treated are reported here.
Groups:
- Total: Total of all reporting groups
Arm/Group | GROUP 1: Cohort 1, Dose Level 1, 3 x10^5 Transduced T Cells/kg (+Or-20%) | GROUP 2: Cohort 1, Dose Level 2, 1x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 3: Cohort 1, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 4: Cohort 1A, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 5: Cohort 1B, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 6: Cohort 2A, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 7: Cohort 2B, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20% | GROUP 8: Cohort 2C, Dose Level 3, 3 x 10^6 Transduced T-cells/kg (+Or- 20%) | Enrolled and Not Assigned to a Treatment Assignment Code; Not Treated | Total
Number analyzed (Participants) | 4 | 4 | 5 | 2 | 1 | 21 | 1 | 1 | 15 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 2 | 0 | 1 | 8 | 1 | 0 | 5 | 18
  Between 18 and 65 years | 3 | 4 | 3 | 2 | 0 | 13 | 0 | 1 | 10 | 36
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.88 (6.06) | 24.75 (3.97) | 19.12 (8.73) | 25.75 (3.45) | 9.7 (0) | 21 (10.86) | 18.2 (0) | 22.6 (0) | 21.75 (10.91) | 20.69 (10.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 2 | 1 | 1 | 9 | 1 | 0 | 6 | 21
  Male | 3 | 4 | 3 | 1 | 0 | 12 | 0 | 1 | 9 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 2 | 0 | 0 | 12 | 0 | 1 | 6 | 24
  Not Hispanic or Latino | 3 | 2 | 3 | 2 | 1 | 9 | 1 | 0 | 7 | 28
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 4
  White | 2 | 2 | 3 | 1 | 1 | 11 | 1 | 1 | 9 | 31
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 1 | 0 | 0 | 6 | 0 | 0 | 3 | 13
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 5 | 2 | 1 | 21 | 1 | 1 | 15 | 54

OUTCOME MEASURES:

1. Primary Outcome: Grades of Toxicity by Type of Toxicity
Description: Safety analyses will consist of tabulations of grades of toxicity by type of toxicity assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0. Grade 1 is mild, Grade 2 is moderate, Grade 3 is severe, Grade 4 is life-threatening, and Grade 5 is death related to adverse event.
Time Frame: From start of lymphodepleting chemotherapy regimen through 30-days after chimeric antigen receptor (CAR) infusion (approximately 5 weeks).
Population: 16/54 participants were not treated including 15 participants that were screen failures. Only grade 3, 4, and 5 toxicities at least possibly related to either research and/or investigational new drug application (IND) will be reported.
Measure: Number; unit: toxicities
Groups:
- GROUP 7: Cohort 2B, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%: Participants who previously received Chimeric Antigen Receptor (CAR) therapy. Dose Level 3, 3 x10^6 transduced T cells/kg (+or-20%Lymphodepleting chemotherapy regimen with Fludarabine and Cyclophosphamide.
  Fludarabine: Fludarabine is administered as an intravenous (IV) infusion in an appropriate solution over 30 minutes. The dose will be based on body surface area (BSA) at 30 mg/m^2/dose on Day -5, -4, -3, -2.
  Cyclophosphamide: Cyclophosphamide will be diluted in an appropriate solution and infused over one hour. The dose will be based on the body surface area (BSA) at 600 mg/m^2/dose after fludarabine infusion on Day -3 & -2.
  Cluster of differentiation 19 (CD19)/cluster of differentiation 22 (CD22)-chimeric antigen receptor (CAR)-transduced T cells at Dose Level 3, 3 x10^6 transduced T cells/kg (+or-20%) infused on Day 0 after lymphodepleting chemotherapy regimen.
Arm/Group | GROUP 1: Cohort 1, Dose Level 1, 3 x10^5 Transduced T Cells/kg (+Or-20%) | GROUP 2: Cohort 1, Dose Level 2, 1x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 3: Cohort 1, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 4: Cohort 1A, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 5: Cohort 1B, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 6: Cohort 2A, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 7: Cohort 2B, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20% | GROUP 8: Cohort 2C, Dose Level 3, 3 x 10^6 Transduced T-cells/kg (+Or- 20%)
Number analyzed (Participants) | 4 | 4 | 4 | 2 | 1 | 21 | 1 | 1
toxicities
  Grade 3 Anemia | 2 | 2 | 1 | 1 | 1 | 13 | 1 | 0
  Grade 3 Febrile neutropenia | 1 | 2 | 1 | 1 | 1 | 13 | 0 | 0
  Grade 3 Sinus tachycardia | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Grade 3 Abdominal pain | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 Diarrhea | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 Gastric hemorrhage | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 3 Fever | 1 | 2 | 0 | 0 | 1 | 3 | 0 | 0
  Grade 3 Cytokine release syndrome | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0
  Grade 3 Immune system disorders, other (GVHD) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 Sepsis | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 3 Alanine aminotransferase | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Grade 3 Aspartate aminotransferase | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
  Grade 3 GGT increased | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 3 Lymphocyte count decreased | 2 | 2 | 4 | 2 | 1 | 13 | 1 | 1
  Grade 3 Neutrophil count decreased | 3 | 2 | 3 | 2 | 0 | 17 | 1 | 1
  Grade 3 Platelet count decreased | 4 | 1 | 0 | 2 | 0 | 8 | 1 | 0
  Grade 3 White blood cell decreased | 3 | 0 | 3 | 2 | 0 | 16 | 1 | 0
  Grade 3 Anorexia | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 Hypertriglyceridemia | 2 | 1 | 0 | 0 | 0 | 3 | 0 | 0
  Grade 3 Hypocalcemia | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 3 Hypokalemia | 0 | 1 | 0 | 0 | 0 | 4 | 0 | 0
  Grade 3 Back pain | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 Myalgia | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Grade 3 Dysphasia | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Grade 3 Encephalopathy | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Grade 3 Headache | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 Nervous system disorder, other (ICANS) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
  Grade 3 Nervous system disorder, other (Neurotoxicity) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Grade 3 Seizure | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
  Grade 3 Hypoxia | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 3 Hypertension | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Grade 3 Hypotension | 0 | 2 | 0 | 1 | 0 | 6 | 0 | 0
  Grade 4 Anemia | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 4 Fibrinogen decreased | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 4 Lymphocyte count decreased | 3 | 3 | 4 | 2 | 1 | 17 | 1 | 1
  Grade 4 Neutrophil count decreased | 3 | 1 | 2 | 2 | 0 | 14 | 1 | 0
  Grade 4 Platelet count decreased | 2 | 1 | 0 | 0 | 1 | 6 | 1 | 0
  Grade 4 White blood cell decreased | 3 | 2 | 0 | 1 | 0 | 10 | 1 | 0
  Grade 4 Hypertriglyceridemia | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 4 Hypokalemia | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

2. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: MTD is defined as the dose level immediately below the level at which the enrollment is stopped due to dose-limiting toxicity (DLT). A DLT is defined as an adverse event that is at least possibly related to the cluster of differentiation 19/cluster of differentiation 22 (CD19/CD22)-chimeric antigen receptor (CAR) T cells with onset within the first 28 days after cell infusion.
Time Frame: First 28 days after cell infusion
Population: 16/54 participants were not treated. Only participants in the dose escalation phase of the study are included in this analysis (Groups 1-5).
Measure: Number; unit: 10^6 CAR T cells/kg
Groups:
- All Participants: All participants who received at least one dose of drug in the dose escalation phase of the study.
Arm/Group | All Participants
Number analyzed (Participants) | 16
10^6 CAR T cells/kg | 3

3. Secondary Outcome: Number of Participants That Have Successful Manufacture of the Targeted Dose Number of Chimeric Antigen Receptor (CAR) Cells
Description: Number of participants that have the targeted dose number of CAR cells successfully manufactured (i.e., number of participants enrolled where the correct number of cells are produces at the dose level that are enrolled) as measured by total number of viable cluster of differentiation 19 (CD19)/cluster of differentiation 22 (CD22) transduced T cells.
Time Frame: CAR infusion (Day 0)
Population: 16/54 participants were not treated.
Measure: Count of Participants; unit: Participants
Groups:
- GROUP 1: Cohort 1, Dose Level 1, 3 x10^5 Transduced T Cells/kg (+Or-20%): Cluster of differentiation 19 (CD19)/cluster of differentiation 22 (CD22)-chimeric antigen receptor (CAR)-transduced T cells Dose Level 1, 3 x10^5 transduced T cells/kg (+or-20%) infused on Day 0 after lymphodepleting chemotherapy regimen.
- GROUP 2: Cohort 1, Dose Level 2, 1x10^6 Transduced T Cells/kg (+Or-20%): Cluster of differentiation 19 (CD19)/cluster of differentiation 22 (CD22)-chimeric antigen receptor (CAR)-transduced T cells at Dose Level 2, 1x10^6 transduced T cells/kg (+or-20%) infused on Day 0 after lymphodepleting chemotherapy regimen.
- GROUP 3: Cohort 1, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%): Cluster of differentiation 19 (CD19)/cluster of differentiation 22 (CD22)-chimeric antigen receptor (CAR)-transduced T cells at Dose Level 3, 3 x10^6 transduced T cells/kg (+or-20%) infused on Day 0 after lymphodepleting chemotherapy regimen.
- GROUP 4: Cohort 1A, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%); GROUP 6: Cohort 2A, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%): Participants who are chimeric antigen receptor (CAR) naïve or CAR pre-treated and received an interval transplant.
  Cluster of differentiation 19 (CD19)/cluster of differentiation 22 (CD22)-chimeric antigen receptor (CAR)-transduced T cells at Dose Level 3, 3 x10^6 transduced T cells/kg (+or-20%) infused on Day 0 after lymphodepleting chemotherapy regimen.
- GROUP 5: Cohort 1B, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%); GROUP 7: Cohort 2B, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%: Participants who previously received Chimeric Antigen Receptor (CAR) therapy. Cluster of differentiation 19 (CD19)/cluster of differentiation 22 (CD22)-chimeric antigen receptor (CAR)-transduced T cells at Dose Level 3, 3 x10^6 transduced T cells/kg (+or-20%) infused on Day 0 after lymphodepleting chemotherapy regimen.
- GROUP 8: Cohort 2C, Dose Level 3, 3 x 10^6 Transduced T-cells/kg (+Or- 20%): Participants with isolated central nervous system (CNS) disease. Cluster of differentiation 19 (CD19)/cluster of differentiation 22 (CD22)-chimeric antigen receptor (CAR)-transduced T cells at Dose Level 3, 3 x10^6 transduced T cells/kg (+or-20%) infused on Day 0 after lymphodepleting chemotherapy regimen.
Arm/Group | GROUP 1: Cohort 1, Dose Level 1, 3 x10^5 Transduced T Cells/kg (+Or-20%) | GROUP 2: Cohort 1, Dose Level 2, 1x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 3: Cohort 1, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 4: Cohort 1A, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 5: Cohort 1B, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 6: Cohort 2A, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 7: Cohort 2B, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20% | GROUP 8: Cohort 2C, Dose Level 3, 3 x 10^6 Transduced T-cells/kg (+Or- 20%)
Number analyzed (Participants) | 4 | 4 | 5 | 2 | 1 | 21 | 1 | 1
Participants | 4 | 4 | 5 | 2 | 1 | 21 | 1 | 1

4. Secondary Outcome: Overall Survival
Description: Overall survival (OS) will be determined as the time from the date of chimeric antigen receptor (CAR) infusion until death.
Time Frame: Number of months from CAR cell infusion until date of death or time of censor (max 66.6 months)
Population: 16/54 participants were not treated.
Measure: Median (Full Range); unit: Months
Groups:
- GROUP 4: Cohort 1A, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%): Patients who are CAR naïve or CAR pre-treated and received an interval transplant.
  Lymphodepleting chemotherapy regimen with Fludarabine and Cyclophosphamide. Fludarabine: Fludarabine is administered as an intravenous (IV) infusion in an appropriate solution over 30 minutes. The dose will be based on body surface area (BSA) at 25 mg/m^2/dose on Day -4, -3, -2.
  Cyclophosphamide: Cyclophosphamide will be diluted in an appropriate solution and infused over one hour. The dose will be based on the body surface area (BSA) at 900 mg/m^2/dose after fludarabine infusion on Day -2.
  Cluster of differentiation 19 (CD19)/cluster of differentiation 22 (CD22)-chimeric antigen receptor (CAR)-transduced T cells at Dose Level 3, 3 x10^6 transduced T cells/kg (+or-20%) infused on Day 0 after lymphodepleting chemotherapy regimen.
Arm/Group | GROUP 1: Cohort 1, Dose Level 1, 3 x10^5 Transduced T Cells/kg (+Or-20%) | GROUP 2: Cohort 1, Dose Level 2, 1x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 3: Cohort 1, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 4: Cohort 1A, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 5: Cohort 1B, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 6: Cohort 2A, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 7: Cohort 2B, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20% | GROUP 8: Cohort 2C, Dose Level 3, 3 x 10^6 Transduced T-cells/kg (+Or- 20%)
Number analyzed (Participants) | 4 | 4 | 4 | 2 | 1 | 21 | 1 | 1
Months | 12.2 [8.9 to 27.8] | 17.8 [10.9 to 68.5] | 45.4 [13 to 66.6] | 15.3 [10.1 to 20.5] | 60 [60 to NA] — The upper end confidence interval cannot be estimated with one participant. | 20.7 [3 to 50.9] | 9.2 [9.2 to NA] — The upper end confidence interval cannot be estimated with one participant. | 8.3 [8.3 to NA] — The upper end confidence interval cannot be estimated with one participant.

5. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is assessed from the date of chimeric antigen receptor (CAR) infusion until the documentation of disease progression or death due to any cause, whichever occurs first. Disease progression was assessed by the Response Criteria Lymphoma and is defined as individual node/lesion must be abnormal with LDI>1.5 cm and increase by ≥50% from product of perpendicular diameters (PPD) nadir and an increase in longest transverse diameter of a lesion (LDI) or shortest axis perpendicular to LDi (SDI) from nadir 0.5 cm for lesions ≤2 cm, 1.0 cm for lesions > 2 cm; and the International Working Group and is defined as worse marrow classification with at least a 50% increase in the percentage of marrow blasts.
Time Frame: Number of months from CAR cell infusion until time of disease progression, death, or date of censor (up to 67 months)
Population: 16/54 participants were not treated.
Measure: Median (Full Range); unit: Months
Groups:
- GROUP 7: Cohort 2B, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%: GROUP 7: Cohort 2B, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20% Participants who previously received Chimeric Antigen Receptor (CAR) therapy.
  Lymphodepleting chemotherapy regimen with Fludarabine and Cyclophosphamide. Fludarabine: Fludarabine is administered as an intravenous (IV) infusion in an appropriate solution over 30 minutes. The dose will be based on body surface area (BSA) at 30 mg/m^2/dose on Day -5, -4, -3, -2.
  Cyclophosphamide: Cyclophosphamide will be diluted in an appropriate solution and infused over one hour. The dose will be based on the body surface area (BSA) at 600 mg/m^2/dose after fludarabine infusion on Day -3 & -2.
  Cluster of differentiation 19 (CD19)/cluster of differentiation 22 (CD22)-chimeric antigen receptor (CAR)-transduced T cells at Dose Level 3, 3 x10^6 transduced T cells/kg (+or-20%) infused on Day 0 after lymphodepleting chemotherapy regimen.
Arm/Group | GROUP 1: Cohort 1, Dose Level 1, 3 x10^5 Transduced T Cells/kg (+Or-20%) | GROUP 2: Cohort 1, Dose Level 2, 1x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 3: Cohort 1, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 4: Cohort 1A, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 5: Cohort 1B, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 6: Cohort 2A, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 7: Cohort 2B, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20% | GROUP 8: Cohort 2C, Dose Level 3, 3 x 10^6 Transduced T-cells/kg (+Or- 20%)
Number analyzed (Participants) | 4 | 4 | 4 | 2 | 1 | 21 | 1 | 1
Months | 6.4 [0.9 to 11.9] | 2.6 [1.0 to 8.6] | 20.1 [0.9 to 66.6] | 5.3 [2.4 to 8.1] | 60 [60 to NA] — The upper end confidence interval cannot be estimated with one participant. | 14.2 [0.9 to 50.9] | 5.7 [5.7 to NA] — The upper end confidence interval cannot be estimated with one participant. | 8.3 [8.3 to NA] — The upper end confidence interval cannot be estimated with one participant.

6. Secondary Outcome: Clinical Activity (Response) in Children and Young Adults With B-cell Acute Lymphoblastic Leukemia (B-ALL), Isolated Central Nervous System (CNS) ALL, or Lymphoma Who Previously Received Chimeric Antigen Receptor (CAR) Therapy and Those That Are CAR Naive
Description: Clinical activity (response) in children (age ≥3 years to 17 years) and young adults (age 18 years to ≤ 39 years) was measured by the Response Criteria Lymphoma. Complete Response (CR) is complete metabolic and/or radiographic response. Partial Response (PR) is partial metabolic response or partial remission. Stable Disease (SD) is no metabolic response or 50% decrease from baseline in the sum of products of diameters (SPD) of up to 6 dominant measurable nodes and extra nodal sites. Progressive Disease (PD) is individual node/lesion must be abnormal with longest transverse diameter of a lesion (LDI) >1.5 cm and increase by ≥50% from product of perpendicular diameters (PPD) nadir and an increase in LDI or shortest axis perpendicular to LDi (SDI) from nadir 0.5 cm for lesions ≤2 cm and/or 1.0 cm for lesions > 2 cm; also assessed by the International Working Group and PD is defined as worse marrow classification with at least a 50% increase in the percentage of marrow blasts.
Time Frame: At Day 28 (+/- 4 days) after CAR cell infusion
Population: 16/54 participants were not treated. Participants treated in Group 1-3 will be excluded from this outcome measure as assignment to CAR naïve versus CAR pre-treated did not occur in the beginning of the trial. The study was not looking at response in children vs young adults separately. It was looking at response in children and young adults only (no adults over 39). Also, it is not powered to look at children and young adults separately.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- GROUP 4:Cohort 1A, CAR Naïve or CAR Pretreated With Interval Hematopoietic Stem Cell Transplantation; GROUP 6:Cohort 2A, CAR Naïve or CAR Pretreated With Interval Hematopoietic Stem Cell Transplantation: Participants who are CAR naïve or CAR pre-treated and received an interval transplant.
  Lymphodepleting chemotherapy regimen with Fludarabine and Cyclophosphamide. Fludarabine: Fludarabine is administered as an intravenous (IV) infusion in an appropriate solution over 30 minutes. The dose will be based on body surface area (BSA) at 25 mg/m^2/dose on Day -4, -3, -2.
  Cyclophosphamide: Cyclophosphamide will be diluted in an appropriate solution and infused over one hour. The dose will be based on the body surface area (BSA) at 900 mg/m^2/dose after fludarabine infusion on Day -2.
  Cluster of differentiation 19 (CD19)/cluster of differentiation 22 (CD22)-chimeric antigen receptor (CAR)-transduced T cells at Dose Level 3, 3 x10^6 transduced T cells/kg (+or-20%) infused on Day 0 after lymphodepleting chemotherapy regimen.
- GROUP 5: Cohort 1B, Previously Received Chimeric Antigen Receptor (CAR) Participants; GROUP 7: Cohort 2B, Previously Received Chimeric Antigen Receptor (CAR): Participants who previously received Chimeric Antigen Receptor (CAR) therapy. Lymphodepleting chemotherapy regimen with Fludarabine and Cyclophosphamide. Fludarabine: Fludarabine is administered as an intravenous (IV) infusion in an appropriate solution over 30 minutes. The dose will be based on body surface area (BSA) at 30 mg/m^2/dose on Day -5, -4, -3, -2.
  Cyclophosphamide: Cyclophosphamide will be diluted in an appropriate solution and infused over one hour. The dose will be based on the body surface area (BSA) at 600 mg/m^2/dose after fludarabine infusion on Day -3 & -2.
  Cluster of differentiation 19 (CD19)/cluster of differentiation 22 (CD22)-chimeric antigen receptor (CAR)-transduced T cells at Dose Level 3, 3 x10^6 transduced T cells/kg (+or-20%) infused on Day 0 after lymphodepleting chemotherapy regimen.
- Group 8:Cohort 2C, CAR Naïve or CAR Pretreated With Previous Hematopoietic Stem Cell Transplantation: Participants with isolated central nervous system (CNS) disease. Lymphodepleting chemotherapy regimen with Fludarabine and Cyclophosphamide. Fludarabine: Fludarabine is administered as an intravenous (IV) infusion in an appropriate solution over 30 minutes. The dose will be based on body surface area (BSA) at 25 mg/m^2/dose on Day -4, -3, -2.
  Cyclophosphamide: Cyclophosphamide will be diluted in an appropriate solution and infused over one hour. The dose will be based on the body surface area (BSA) at 900 mg/m^2/dose after fludarabine infusion on Day -2.
  Cluster of differentiation 19 (CD19)/cluster of differentiation 22 (CD22)-chimeric antigen receptor (CAR)-transduced T cells at Dose Level 3, 3 x10^6 transduced T cells/kg (+or-20%) infused on Day 0 after lymphodepleting chemotherapy regimen.
Arm/Group | GROUP 4:Cohort 1A, CAR Naïve or CAR Pretreated With Interval Hematopoietic Stem Cell Transplantation | GROUP 5: Cohort 1B, Previously Received Chimeric Antigen Receptor (CAR) Participants | GROUP 6:Cohort 2A, CAR Naïve or CAR Pretreated With Interval Hematopoietic Stem Cell Transplantation | GROUP 7: Cohort 2B, Previously Received Chimeric Antigen Receptor (CAR) | Group 8:Cohort 2C, CAR Naïve or CAR Pretreated With Previous Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 2 | 1 | 21 | 1 | 1
percentage of participants
  CR in children and young adults | 50 [2.6 to 97.4] | 100 [5.1 to 100] | 90.5 [71.1 to 98.3] | 100 [5.1 to 100] | 100 [5.1 to 100]
  PR in children and young adults | 50 [2.6 to 97.4] | 0 [0 to 94.9] | 0 [0 to 15.5] | 0 [0 to 94.9] | 0 [0 to 94.9]
  SD in children and young adults | 0 [0 to 82.2] | 0 [0 to 94.9] | 0 [0 to 15.5] | 0 [0 to 94.9] | 0 [0 to 94.9]
  PD in children and young adults | 0 [0 to 82.2] | 0 [0 to 94.9] | 9.5 [1.7 to 28.9] | 0 [0 to 94.9] | 0 [0 to 94.9]

7. Other Pre Specified Outcome: Number of Participants With a Dose-limiting Toxicity (DLT)
Description: A DLT is defined as an adverse event that is at least possibly related to the cluster of differentiation 19/cluster of differentiation 22 (CD19/CD22)-chimeric antigen receptor (CAR) T cells with onset within the first 28 days after cell infusion.
Time Frame: First 28 days
Population: 16/54 participants were not treated.
Measure: Count of Participants; unit: Participants
Groups:
- GROUP 8: Cohort 2C, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or- 20%): Participants with isolated central nervous system (CNS) disease. Lymphodepleting chemotherapy regimen with Fludarabine and Cyclophosphamide. Fludarabine: Fludarabine is administered as an intravenous (IV) infusion in an appropriate solution over 30 minutes. The dose will be based on body surface area (BSA) at 25 mg/m^2/dose on Day -4, -3, -2.
  Cyclophosphamide: Cyclophosphamide will be diluted in an appropriate solution and infused over one hour. The dose will be based on the body surface area (BSA) at 900 mg/m^2/dose after fludarabine infusion on Day -2.
  Cluster of differentiation 19 (CD19)/cluster of differentiation 22 (CD22)-chimeric antigen receptor (CAR)-transduced T cells at Dose Level 3, 3 x10^6 transduced T cells/kg (+or-20%) infused on Day 0 after lymphodepleting chemotherapy regimen.
Arm/Group | GROUP 1: Cohort 1, Dose Level 1, 3 x10^5 Transduced T Cells/kg (+Or-20%) | GROUP 2: Cohort 1, Dose Level 2, 1x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 3: Cohort 1, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 4: Cohort 1A, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 5: Cohort 1B, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 6: Cohort 2A, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 7: Cohort 2B, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20% | GROUP 8: Cohort 2C, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or- 20%)
Number analyzed (Participants) | 4 | 4 | 4 | 2 | 1 | 21 | 1 | 1
Participants | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0

8. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0).
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Adverse Events were monitored/assessed from the first study intervention, Study Day -4, through day 30 after the study agent (s) was/were administered, an average of 5 weeks.
Population: 16/54 participants were not treated.
Measure: Count of Participants; unit: Participants
Arm/Group | GROUP 1: Cohort 1, Dose Level 1, 3 x10^5 Transduced T Cells/kg (+Or-20%) | GROUP 2: Cohort 1, Dose Level 2, 1x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 3: Cohort 1, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 4: Cohort 1A, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 5: Cohort 1B, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 6: Cohort 2A, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 7: Cohort 2B, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20% | Group 8:Cohort 2C, CAR Naïve or CAR Pretreated With Previous Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 4 | 4 | 4 | 2 | 1 | 21 | 1 | 1
Participants | 4 | 4 | 4 | 2 | 1 | 21 | 1 | 1

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored/assessed an average of 35 days. Adverse Events were monitored/assessed from the first study intervention (Study Day -4, through day 30 after the study agent (s) was/were administered) in any cycle, an average of 5 weeks.
Description: 16/54 participants were not treated.
Arm/Group | GROUP 1: Cohort 1, Dose Level 1, 3 x10^5 Transduced T Cells/kg (+Or-20%) | GROUP 2: Cohort 1, Dose Level 2, 1x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 3: Cohort 1, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 4: Cohort 1A, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 5: Cohort 1B, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 6: Cohort 2A, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) | GROUP 7: Cohort 2B, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20% | Group 8:Cohort 2C, CAR Naïve or CAR Pretreated With Previous Hematopoietic Stem Cell Transplantation
All-Cause Mortality (participants affected / at risk) | 4/4 | 3/4 | 2/4 | 2/2 | 0/1 | 8/21 | 1/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 2/4 | 2/4 | 0/4 | 2/2 | 1/1 | 7/21 | 0/1 | 1/1
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 4/4 | 2/2 | 1/1 | 21/21 | 1/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GROUP 1: Cohort 1, Dose Level 1, 3 x10^5 Transduced T Cells/kg (+Or-20%) (N=4) | GROUP 2: Cohort 1, Dose Level 2, 1x10^6 Transduced T Cells/kg (+Or-20%) (N=4) | GROUP 3: Cohort 1, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) (N=4) | GROUP 4: Cohort 1A, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) (N=2) | GROUP 5: Cohort 1B, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) (N=1) | GROUP 6: Cohort 2A, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) (N=21) | GROUP 7: Cohort 2B, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20% (N=1) | Group 8:Cohort 2C, CAR Naïve or CAR Pretreated With Previous Hematopoietic Stem Cell Transplantation (N=1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GGT increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Immune system disorders - Other, GVHD (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, COVID-19(omicron strain is >90%) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorders - Other, (Neurotoxicity) (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders - Other, ICANS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorders - Other, ICANS level grade 3 CTCAE v5 grade 3 (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GROUP 1: Cohort 1, Dose Level 1, 3 x10^5 Transduced T Cells/kg (+Or-20%) (N=4) | GROUP 2: Cohort 1, Dose Level 2, 1x10^6 Transduced T Cells/kg (+Or-20%) (N=4) | GROUP 3: Cohort 1, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) (N=4) | GROUP 4: Cohort 1A, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) (N=2) | GROUP 5: Cohort 1B, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) (N=1) | GROUP 6: Cohort 2A, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20%) (N=21) | GROUP 7: Cohort 2B, Dose Level 3, 3 x10^6 Transduced T Cells/kg (+Or-20% (N=1) | Group 8:Cohort 2C, CAR Naïve or CAR Pretreated With Previous Hematopoietic Stem Cell Transplantation (N=1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 2 (3) | 2 (6) | 2 (4) | 1 (1) | 10 (17) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (2) | 1 (1) | 2 (4) | 1 (3) | 1 (1) | 9 (12) | 1 (4) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (15) | 3 (8) | 2 (2) | 2 (4) | 1 (2) | 9 (17) | 0 (0) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (2) | 2 (4) | 2 (2) | 0 (0) | 0 (0) | 5 (7) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 4 (19) | 4 (7) | 4 (8) | 2 (13) | 1 (11) | 19 (116) | 1 (8) | 1 (3)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 2 (3) | 3 (8) | 2 (5) | 0 (0) | 13 (16) | 1 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2) | 2 (3) | 2 (4) | 1 (3) | 10 (13) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (6) | 2 (7) | 0 (0) | 2 (9) | 1 (6) | 13 (37) | 1 (1) | 1 (4)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 3 (3) | 1 (2) | 1 (3) | 13 (17) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other, specify: Inguinal lymph node enlarged on L (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bicarbonate decreased (Investigations) | 0 (0) | 1 (2) | 3 (12) | 2 (6) | 1 (1) | 13 (31) | 0 (0) | 1 (4)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 1 (2) | 0 (0) | 10 (29) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (3) | 1 (3) | 1 (1) | 2 (6) | 1 (1) | 15 (30) | 1 (1) | 1 (1)
Blood prolactin abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 9 (13) | 1 (1) | 0 (0)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CPK increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3)
Cardiac disorders - Other, specify: Grade II/VI systolic ejection murmur at LSB (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac disorders - Other, specify: Hypokinesia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 2 (3) | 2 (3) | 3 (3) | 1 (2) | 0 (0) | 8 (9) | 1 (1) | 0 (0)
Cholesterol high (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 7 (8) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 10 (13) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 6 (10) | 0 (0) | 0 (0)
Cushingoid (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 16 (19) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (10) | 1 (1) | 10 (12) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 7 (10) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (6) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 9 (11) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (3) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema face (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 7 (8) | 0 (0) | 0 (0)
Edema trunk (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Eye disorders - Other, specify: Irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye disorders - Other, specify: Right visual field cut, (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye disorders - Other, specify: corneal abrasion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 4 (6) | 1 (1) | 2 (3) | 0 (0) | 14 (25) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (4) | 1 (2) | 1 (1) | 1 (1) | 13 (17) | 0 (0) | 0 (0)
Fecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 2 (10) | 2 (8) | 2 (6) | 2 (6) | 1 (4) | 17 (53) | 0 (0) | 0 (0)
Fibrinogen decreased (Investigations) | 2 (4) | 1 (2) | 0 (0) | 1 (1) | 1 (2) | 9 (25) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GGT increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (7) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify: Mucosal colored protrusion in mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Glucosuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haptoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 4 (9) | 3 (9) | 2 (12) | 1 (2) | 17 (46) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatobiliary disorders - Other, specify: Gallbladder wall/periportal edema (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (6) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (3) | 3 (14) | 4 (17) | 2 (18) | 1 (1) | 16 (61) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 (0) | 4 (16) | 4 (9) | 1 (1) | 0 (0) | 9 (18) | 1 (5) | 0 (0)
Hypertension (Vascular disorders) | 2 (4) | 1 (1) | 0 (0) | 1 (1) | 1 (6) | 2 (2) | 0 (0) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 3 (12) | 3 (21) | 2 (6) | 2 (9) | 1 (3) | 16 (49) | 0 (0) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 8 (20) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (9) | 2 (5) | 1 (2) | 2 (14) | 1 (4) | 18 (48) | 1 (1) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 2 (4) | 1 (1) | 2 (5) | 1 (1) | 11 (25) | 1 (1) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (8) | 4 (15) | 0 (0) | 1 (7) | 1 (3) | 18 (48) | 1 (2) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 9 (19) | 1 (1) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (4) | 1 (2) | 2 (5) | 2 (10) | 1 (1) | 15 (31) | 1 (2) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (4) | 1 (4) | 13 (30) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 3 (3) | 1 (1) | 2 (4) | 0 (0) | 9 (14) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
INR increased (Investigations) | 3 (4) | 3 (6) | 2 (2) | 1 (2) | 0 (0) | 5 (9) | 0 (0) | 0 (0)
Infections and infestations - Other, specify: Bacteroides fragilis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify: C.difficile (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, specify: CMV (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify: COVID (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Infections and infestations - Other, specify: Coronavirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, specify: HSV (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, specify: Norovirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, specify: Rhino/enterovirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, specify: Staph blepharitis Rt Eye (Ophth note) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify: Staphylococcus epidermidis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify: gram negative rod (E. Coli) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (3) | 2 (4) | 1 (1) | 1 (1) | 1 (1) | 4 (5) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Localized edema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (19) | 3 (11) | 4 (41) | 2 (33) | 1 (2) | 21 (123) | 1 (10) | 1 (8)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Movements involuntary (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify: Wrist joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (4) | 1 (3) | 0 (0) | 7 (14) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (5) | 4 (10) | 2 (5) | 1 (2) | 17 (33) | 0 (0) | 1 (1)
Neck edema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (2) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (36) | 2 (15) | 4 (37) | 2 (26) | 0 (0) | 21 (137) | 1 (5) | 1 (3)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 3 (9) | 4 (8) | 2 (8) | 0 (0) | 16 (29) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 11 (15) | 1 (2) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 4 (34) | 4 (9) | 4 (10) | 2 (13) | 1 (4) | 19 (66) | 1 (7) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (5) | 2 (3) | 2 (3) | 0 (0) | 3 (5) | 0 (0) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (5) | 1 (1) | 1 (1) | 0 (0) | 3 (6) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify: Lung nodule (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scrotal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 2 (3) | 3 (5) | 2 (6) | 1 (3) | 16 (27) | 1 (2) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 4 (8) | 4 (5) | 4 (8) | 2 (4) | 0 (0) | 10 (16) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendon reflex decreased (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (4) | 3 (4) | 3 (6) | 1 (2) | 1 (2) | 13 (23) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 3 (25) | 3 (12) | 4 (41) | 2 (27) | 0 (0) | 20 (151) | 1 (7) | 1 (4)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flu-like symptoms (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune system disorders, other GVHD (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2024-11-19): https://cdn.clinicaltrials.gov/large-docs/93/NCT03448393/Prot_SAP_000.pdf
  • Informed Consent Form: Cohort Standard, Parental or Guardian Permission for Minor (2024-06-18): https://cdn.clinicaltrials.gov/large-docs/93/NCT03448393/ICF_001.pdf
  • Informed Consent Form: Cohort Assent Minors, 12-17 Years Old (2024-06-18): https://cdn.clinicaltrials.gov/large-docs/93/NCT03448393/ICF_002.pdf